CLINICAL TRIAL: NCT05903833
Title: Pembrolizumab in Combination With Lenvatinib in Pts With Recurrent, Persistent, Metastatic or Locally Advanced Vulvar Cancer Not Amenable to Curative Surgery or Radiotherapy
Brief Title: Pembrolizumab Combination With Lenvatinib in Pts With Recurrent,Persistent,Metastatic or Locally Advanced Vulvar Cancer Not Amenable to Curative Surgery or Radiotherapy
Acronym: PIERCE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AGO Research GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGO-Vulva 1; 2024-515646-16-00 (Other: EU CT Number)
Record Dates: First submitted 2023-05-11; First posted 2023-06-15 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Vulvar Cancer; Persistent Vulvar Cancer; Metastatic Vulva Cancer; Locally Advanced Vulvar Cancer
Keywords: Advanced vulvar cancer; Recurrent vulvar cancer; Persistent vulvar canser; Metastatic vulvar cancer; Locally advanced vulvar cancer; Pembrolizumab; Lenvatinib
MeSH Terms: conditions — Vulvar Neoplasms | interventions — pembrolizumab; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment allocation (Experimental): Administration of pembrolizumab 400 mg Q6W in combination with lenvatinib 20 mg QD
  Interventions: Drug: Pembrolizumab; Drug: Lenvatinib

INTERVENTIONS:
Drug: Pembrolizumab — 400 mg Q6W
Drug: Lenvatinib — 20 mg QD

SUMMARY:
Evaluation of efficacy and safety of pembrolizumab in combination with lenvatinib in patients with recurrent, persistent, metastatic or locally advanced vulva cancer.

DETAILED DESCRIPTION:
A multicenter, single-arm phase II, open-label study, to evaluate the efficacy and safety of pembrolizumab 400 mg Q6W in combination with lenvatinib 20 mg QD in patients with recurrent, persistent, metastatic or locally advanced VSCC not amenable to salvage surgery or definitive (chemo)radiation.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent obtained prior to initiation of any study-specific procedures and treatment as confirmation of the patients awareness and willingness to comply with the study requirements.
2. Female patients who are at least 18 years of age on the day signing informed consent
3. Histologically confirmed locally advanced, recurrent, persistent and/or metastatic VSCC not amenable for salvage surgery or definitive (chemo)radiation (additive palliative radiotherapy for symptom control is allowed)
4. ≤2 previous lines of chemotherapy for recurrent or metastatic disease
5. Measurable disease (investigator assessed RECIST 1.1). Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
6. Have an eastern cooperative oncology group (ECOG) performance status of 0-1. Evaluation of ECOG is to be performed within 7 days prior to the first dose of study intervention.
7. No pregnancy (as documented by a positive beta-human chorionic gonadotropin [ß-hCG] or human chorionic gonadotropin [hCG]) test with a minimum sensitivity of 25 IU/L or equivalent units of ß-hCG [or hCG]), no breastfeeding, and at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 4 OR
   2. A WOCBP who agrees to follow the contraception and pregnancy testing recommendations for investigational medicinal products (IMPs) with demonstrated or suspected human teratogenicity/ fetotoxicity in early pregnancy of the CTFG-guideline in Appendix 4 during the treatment period and for at least 4 months (corresponding to time needed to eliminate pembrolizumab) after the last dose of study treatment. In addition to the described highly effective oral/transdermal contraception methods a barrier method must be used.

   A WOCBP should not become pregnant during the treatment and for at least four months.
8. Available archival tumor tissue sample and/or newly obtained core or excisional biopsy of a tumor lesion ideally not previously irradiated. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides.
9. Adequate organ function as defined in Table 3 of study protocol. Specimens must be collected within 10 days prior to the start of study treatment.

Exclusion Criteria:

1. Non squamous cell histology
2. Contraindications regarding treatment with pembrolizumab:

   allergy or hypersensitivity to pembrolizumab or one of the components.
3. Contraindications regarding treatment with lenvatinib: allergy or hypersensitivity to lenvatinib or one of the components or:

   1. Pre-existing ≥Grade 3 gastrointestinal or nongastrointestinal fistula
   2. Radiographic evidence of major blood vessel infiltration
4. Bradyarrhythmia
5. Arterial dissection/aneurysm
6. Long QT Syndrome
7. Significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina, myocardial infarction or stroke within 12 months of the first dose of study drug, or cardiac arrhythmia requiring medical treatment at screening.
8. History or evidence of major thrombotic (e.g. symptomatic pulmonary embolism) or hemorrhagic disorders within 6 months prior to day 1, cycle 1. The degree of tumor invasion/infiltration of major blood vessels (e.g. carotid artery) should be considered because of the potential risk of severe haemorrhage associated with tumor shrinkage/necrosis following lenvatinib therapy.
9. Allogenic tissue/solid organ transplant.
10. Diagnosis of immunodeficiency
11. Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
12. History of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years (time requirement does not apply for definitively treated early endometrial cancer (FIGO IA/B), in-situ carcinomas [e.g. breast, cervix, bladder], or basal or squamous cell carcinoma of the skin).
13. Gastrointestinal malabsorption, gastrointestinal anastomosis, or any other condition that might affect the absorption of lenvatinib.
14. Active CNS metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
15. History of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
16. Active infection requiring systematic therapy.
17. Has active hemoptysis within 3 weeks prior to the first dose of study intervention or tumor bleeding within 2 weeks prior randomization.
18. Known history of Human Immunodeficiency Virus (HIV) infection
19. History of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection.
20. Known history of active TB (Bacillus tuberculosis).
21. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
22. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
23. Pregnancy
24. Breastfeeding Prior/ Concomitant Therapy
25. Prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or coinhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
26. Systemic use of corticosteroids or immunosuppressive drugs within 7 days prior start of study treatment (see EC 11.)

    * Systemic corticosteroids (at dose higher than 10 mg/day equivalent prednisone); if systemic corticoid use, corticoid must be stopped at least 7 days before study treatment start
    * Interferons
    * Interleukins
    * Live vaccine

    Note: Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster, yellow fever, rabies, BCG, and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed as other killed vaccines, if done at least 2 weeks prior the first dose of study drug; however, intranasal influenza vaccines (e.g. FluMist®) are live attenuated vaccines and are not allowed.
27. Antiarrhythmics of classes Ia and III and other QT-interval prolongation drugs
28. Prior systemic anti-cancer therapy including investigational agents within 4 weeks [could consider shorter interval for kinase inhibitors or other short half-life drugs] prior to allocation.
29. Prior radiotherapy within 2 weeks of start of study intervention. Patients must have recovered from radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
30. Not recovered adequately from any toxicity from other anticancer treatment regimens and/or complications from major surgery prior to starting therapy. Note: Withhold lenvatinib for at least 1 week prior to elective surgery. Do not administer for at least 2 weeks following major surgery and until adequate wound healing.
31. Administration of a live, attenuated vaccine within 30 days prior first dose of study drug. Diagnostic Assessments
32. Uncontrolled blood pressure (Systolic BP >140 mmHg or diastolic BP >90 mmHg) in spite of an optimized regimen of antihypertensive medication.
33. Change of anti-HTN (hypertension) medical regimen within 1 week prior to randomization
34. Prolongation of corrected QT interval (QTc interval) >480 ms
35. Left ventricular ejection fraction (LVEF) below the institutional normal range as determined by multigated acquisition scan (MUGA) or echocardiogram (ECHO).
36. Electrolyte abnormalities that have not been corrected.
37. Subjects having >1+ proteinuria on urine dipstick testing unless a 24-hour urine collection for quantitative assessment indicates that the urine protein is <1 g/24 hours. Prior/Concurrent Study Experience
38. Prior enrolment on a clinical study evaluating pembrolizumab and lenvatinib for a carcinoma, regardless of treatment received.
39. Currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention. Note: Patients who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2029-10-30 (Estimated)

PRIMARY OUTCOMES:
ORR within 24 weeks | 24 weeks
  ORR will be defined as the proportion of patients with PR or CR within 24 weeks starting with the first study treatment. Tumor responses will be assessed by the investigator per Response Evaluation Criteria in Solid Tumors (RECIST 1.1)

SECONDARY OUTCOMES:
Evaluate the efficacy of lenvatinib + pembrolizumab in terms of overall ORR | From date of starting study treatment until the date of first documented progression or date of death from any cause, whichever occurs earlier, assessed up to 40 months
  Overall ORR
Evaluate the efficacy of lenvatinib + pembrolizumab in terms of disease control rate (DCR) | For 8 weeks
  DCR will be defined as the proportion of patients with PR, CR or stable disease (SD)
Evaluate the efficacy of lenvatinib + pembrolizumab in terms of duration of response (DOR) | Time from response until first progression or death, whichever occurs first, assessed up to 40 months
  DOR will be defined as time from response until first progression or death, whichever occurs first
Evaluate the efficacy of lenvatinib + pembrolizumab in terms of overall survival (OS) | Time from date of starting study treatment to death, assessed up to 40 months
  OS will be defined as the time from date of starting study treatment to death.
Evaluate the efficacy of lenvatinib + pembrolizumab in terms of progression free survival (PFS) | Time from starting study treatment to progressive disease or death, whichever occurs first, assessed up to 40 months
  PFS will be defined as the time from starting study treatment to progressive disease (PD) or death, whichever occurs first
Evaluate the efficacy of lenvatinib + pembrolizumab in terms of time to first subsequent therapy (TFST) | The time from date of starting study treatment until the start of the first subsequent therapy or death whichever occurs first, assessed up to 40 months
  • TFST will be defined as the time from date of starting study treatment until the start of the first subsequent therapy or death whichever occurs first.
Evaluate the efficacy of lenvatinib + pembrolizumab in terms of time to second subsequent therapy (TSST) | Time from date of starting study treatment until the start of second subsequent treatment or death whichever occurs first, assessed up to 40 motnhs
  • TSST will be defined as the time from date of starting study treatment until the start of second subsequent treatment or death whichever occurs first.
Patient reported outcomes (QLQ) | Assessed frequently during the trial up to 40 months
  Quality of life is measured by patient reported outcome instruments EORTC QLQ C-30 to evaluate the efficacy of combination of lenvatinib and pembrolizumab
Patient reported outcomes (QLQ) | Assessed frequently during the trial up to 40 months
  Quality of life is measured by patient reported outcome instruments EORTC QLQ VU34 to evaluate the efficacy of combination of lenvatinib and pembrolizumab
Number of participants with treatment-related adverse events (AE) and/or serious adverse events (SAEs) and/or AEs that led to premature withdrawal of trial treatment and/or interruptions/dose modifications | At every visit during the trial up to safety follow, thereafter up to 120 days after administration of last dose of study medication
  Graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, to evaluate the safety and tolerability of the combination of lenvatinib and pembrolizumab

CONTACTS AND LOCATIONS:
Overall Officials: Linn Wölber, MD PhD, Principal Investigator — UKE Hamburg
Locations (15):
- Germany (15):
  - Universitätsklinikum Augsburg, Augsburg
  - Hochtaunus-Kliniken Bad Homburg, Bad Homburg
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - KEM Kliniken Essen-Mitte, Essen
  - Universitätsklinikum Essen, Essen
  - Universitätsmedizin Göttingen, Göttingen
  - University Hospital Hamburg, Hamburg
  - Klinikum Hanau GmbH, Hanau
  - ZAGO - Zentrum für ambulante gynäkologische Onkologie, Krefeld
  - Universitätsmedizin Mainz, Mainz
  - Universitätsklinikum Mannheim, Manheim
  - Klinikum der Universität München, LMU, München
  - Universitätsklinikum Münster, Münster
  - University Hospital, Tübingen

REFERENCES:
- See also: Homepage of AGO Research GmbH — http://www.ago-ovar.de/